CLINICAL TRIAL: NCT06650826
Title: The APIT Study: Prospective Observational Study of the Incidence of Anti-platelet Factor 4 Antibodies in Suspected Immune-associated Arterial and/or Venous Thrombosis
Brief Title: Study Regarding the Incidence of Anti-platelet Factor 4-antibodies in Patients Aged 18 to 60 Years With Spontaneous or Infection- or Vaccine-associated or Recurrent Venous and/or Arterial Thrombosis
Status: Recruiting | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, Clinical Professor, Cardioangiologisches Centrum Bethanien
Other Study IDs: APIT
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Arterial or Venous Thrombosis
Keywords: Anti-PF4 antibodies; infections; vaccination
MeSH Terms: conditions — Venous Thrombosis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples kept at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Spontaneous arterial and/or venous thrombosis: Patients with spontaneous arterial and/or venous thrombosis
  Interventions: Diagnostic Test: Determination of anti-platelet factor 4 antibodies in the blood
- Infection-associated arterial and/or venous thrombosis: Patients with infection-associated arterial and/or venous thrombosis
  Interventions: Diagnostic Test: Determination of anti-platelet factor 4 antibodies in the blood
- Vaccine-associated arterial and/or venous thrombosis: Patients with vaccine-associated arterial and/or venous thrombosis
  Interventions: Diagnostic Test: Determination of anti-platelet factor 4 antibodies in the blood
- Recurrent arterial and/or venous thrombosis despite anticoagulant therapy: Patients with recurrent arterial and/or venous thrombosis despite anticoagulant therapy
  Interventions: Diagnostic Test: Determination of anti-platelet factor 4 antibodies in the blood

INTERVENTIONS:
Diagnostic Test: Determination of anti-platelet factor 4 antibodies in the blood — The anti-platelet factor 4 antibodies in the blood are determined using latex agglutination and the chemiluminescence method in the coagulation laboratory of the CCB MVZ laboratory. In addition, the platelet factor 4-induced platelet activation test (PIPA test) and the heparin-induced platelet activation test (HIPA test) as well as an ELISA-based platelet factor 4 IgG antibody test (Prof. Greinacher, Greifswald University Hospital) will be performed as part of the routine work up.
  In addition a new assay for heparin-independent anti-PF4 antibody detection provided by the company Werfen using chemiluminescence will be performed.

SUMMARY:
Prospective investigation of the incidence of anti-platelet factor 4 antibodies in suspected immune-associated arterial and/or venous thrombosis

DETAILED DESCRIPTION:
Patients with venous and/or arterial thrombosis aged 18 to 60 years are included.Thromboses should have occurred spontaneously or within 30 days after an infection or vaccination. In addition, patients with recurrent thrombosis, despite anticoagulation, are also included in the study. The primary aim of the study is to determine the incidence of anti-platelet factor 4 antibodies in relation to venous and/or arterial thrombosis. For this purpose, we will take a blood sample from the patients within 120 days of the occurrence of the thrombosis.

As a secondary objective, platelet count, D-dimer and results of a thrombophilia screening as well as thrombosis localization are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years
* Written informed consent of the patient
* Spontaneous arterial and/or venous thrombosis
* infection-associated arterial and/or venous thrombosis within 30 days of infection
* Vaccine-associated arterial and/or venous thrombosis within 30 days of vaccination
* Recurrent arterial or venous thrombosis despite anticoagulant therapy

Exclusion Criteria:

* Lack of consent of the patient
* Risk-associated venous thromboses (e.g. following surgery, immobilization, plaster cast, fractures or sprains)
* Risk-associated arterial thromboses (in the presence of vascular risk factors such e.g. diabetes mellitus, hypercholesterolemia, hypertension, nicotine abuse)
* Thromboses more than 120 days old at the time of blood sampling

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with venous and/or arterial thromboses that occur spontaneously, in association with infections or vaccinations or recurrently and are not associated with the presence of typical risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Presence of anti-platelet factor 4 antibodies in temporal connection with the occurrence of arterial and/or venous thrombosis | Day 1
  Presence of anti-platelet factor 4 antibodies in temporal connection with the occurrence of arterial and/or venous thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Professor, Principal Investigator — Cardioangiologisches Zentrum Bethanien
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum der Charite (DHZC), Berlin
  - Cardioangiologisches Zentrum Bethanien (CCB), Frankfurt am Main

IPD SHARING:
Plan to Share IPD: No